CLINICAL TRIAL: NCT04950322
Title: A Randomized, Double-Blind, Multi-Center, Phase III Clinical Study of SHR-1701 Plus Chemotherapy Versus Placebo Plus Chemotherapy as Treatment in Patients With Previously Untreated, Advanced or Metastatic Gastric or Gastroesophageal Junction Cancer
Brief Title: A Trial of SHR1701 Plus Chemotherapy in Patients With Gastric or Gastroesophageal Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1701-III-307
Record Dates: First submitted 2021-06-29; First posted 2021-07-06 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Gastric or Gastroesophageal Junction Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-1701、CAPOX
- Treatment group B (Placebo Comparator)
  Interventions: Drug: Placebo、CAPOX

INTERVENTIONS:
Drug: SHR-1701、CAPOX — SHR-1701 with CAPOX (CAPOX:Oxaliplatin,Capecitabine)
  Arms: Treatment group A
Drug: Placebo、CAPOX — Placebo with CAPOX (CAPOX:Oxaliplatin,Capecitabine)
  Arms: Treatment group B

SUMMARY:
This study is a randomized, Double-Blind, multi-center Phase III clinical study, aimed to evaluate the efficacy and safety of SHR1701 combined with chemotherapy in the treatment of Previously Untreated, Advanced or Metastatic Gastric or Gastroesophageal Junction Cancer. For Part 1 study，the tolerability of SHR-1701 will be evaluated and determine the recommended dose for Part 2.For Part 2 study, all enrolled patients will be randomized to 2 groups and continuously treated until the end criteria of treatment was met.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of locally advanced unresectable or metastatic gastric or gastroesophageal junction (GEJ)adenocarcinoma.
2. HER2 overexpression or amplification negative.
3. Female or male, 18 years of age or above.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
5. Patients who are willing and able to provide the signed informed consent form, willing and able to comply with all the scheduled visits, study treatment, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Squamous cell carcinoma, undifferentiated carcinoma, or other histological types of gastric cancer.
2. Presence of inadequately treated CNS metastases, or uncontrolled or symptomatic active CNS metastases ，leptomeningeal disease, and/or rapid progression.
3. Presence of uncontrolled pleural effusion or ascites despite puncture drainage within 14 days prior to randomization.
4. More than 20% weight loss within 2 months prior to randomization.
5. Diagnosed with other malignant tumors within 5 years prior to enrollment.
6. Presence of any active, known or suspected autoimmune disease.
7. Prior treatment with TGF-β inhibitor, anti-PD-1/PD-L1 antibodies, anti-PD-L2 antibodies, anti-CD137 antibodies, anti-CTLA-4 antibodies, or other drugs/antibodies.
8. Severe, unhealed, or dehisced wounds and active ulcers or untreated fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
AEs and SAEs in part 1 study | up to 2 years
  The number and proportion of subjects with dose limiting toxicity. The safety endpoints, including incidence and severity of adverse events (AEs) and serious adverse events (SAEs).
Overall survival in subjects with PD-L1 CPS ≥ 5 in part 2 study | up to 3 years
OS in all subjects in part 2 study | up to 3 years
  Overall survival (OS)

SECONDARY OUTCOMES:
ORR in part 1 study | up to 2 years
  Objective response rate (ORR) as assessed by the investigator per RECIST 1.1
DCR in part 1 study | up to 2 years
  Disease control rate (DCR) as assessed by the investigator per RECIST 1.1
PFS in part 1 study | up to 2 years
  Progression free survival (PFS) as assessed by the investigator per RECIST 1.1
DoR in part 1 study | up to 2 years
  Duration of response (DoR) as assessed by the investigator per RECIST 1.1
OS in part 1 study | up to 3 years
  Overall survival (OS)
PFS in part 2 study | up to 3 years
  PFS in subjects with PD-L1 CPS ≥5 and in all subjects as assessed by BICR per RECIST 1.1
ORR in part 2 study | up to 2 years
  ORR in subjects with PD-L1 CPS ≥5 and in all subjects as assessed by BICR per RECIST 1.1
DCR in part 2 study | up to 2 years
  DCR in subjects with PD-L1 CPS ≥5 and in all subjects as assessed by BICR per RECIST 1.1
DoR in part2 study | up to 2 years
  DoR in subjects with PD-L1 CPS ≥5 and in all subjects as assessed by BICR per RECIST 1.1
PFS in subjects with PD-L1 CPS ≥5 and in all subjects as assessed by investigator as per RECIST 1.1 | up to 2 years
ORR in part 2 study | up to 2 years
  ORR in subjects with PD-L1 CPS ≥5 and in all subjects as assessed by investigator per RECIST 1.1
DCR in part 2 study | up to 2 years
  DCR in subjects with PD-L1 CPS ≥5 and in all subjects as assessed by investigator per RECIST 1.1
DoR in part 2 study | up to 2 years
  DoR in subjects with PD-L1 CPS ≥5 and in all subjects as assessed by investigator per RECIST 1.1
AEs and SAEs in part 2 study | up to 2 years
  Safety endpoints, including incidence and severity of AEs and SAEs as per NCI-CTCAE v5.0 criteria
EORTC QLQ-C30 score | up to 2 years
EORTC QLQ-STO22 score | up to 2 years
EQ-5D-5L score | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided